CLINICAL TRIAL: NCT02564237
Title: A Phase I, Randomized, Observer-blind, Comparator-controlled, Study of the Safety and Immunogenicity of StreptAnova™ Vaccine in Healthy Adults Age ≥ 18 - 50 Years
Brief Title: A Controlled Study to Evaluate the Safety and Immunogenicity of StreptAnova™ in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Shelly A. McNeil, Professor and Head, Division of Infectious Diseases, Dept Medicine, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PE1201
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Group A streptococcal
MeSH Terms: interventions — Vaccines; Hepatitis B Vaccines; Hepatitis A Vaccines; Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: StreptAnova™ (Experimental): Three (3) 0.6 mL doses (600 µg protein) of StreptAnova™ (Group A streptococcal (GAS) vaccine) will be will be administered on days 0, 30 and 180.
  Interventions: Biological: StreptAnova™ (Group A streptococcal (GAS) vaccine)
- Group 2: Comparator (Active Comparator): Three (3) 0.5 mL doses of comparator (Hepatitis B vaccine, Hepatitis A vaccine, OR Human Papillomavirus vaccine) will be administered on days 0, 30 and 180.
  Interventions: Biological: Hepatitis B vaccine; Biological: Hepatitis A vaccine; Biological: Human Papillomavirus vaccine

INTERVENTIONS:
Biological: StreptAnova™ (Group A streptococcal (GAS) vaccine) — StreptAnova™ vaccine - 30-valent plus Spa group A Streptococcal vaccine
  Arms: Group 1: StreptAnova™
Biological: Hepatitis B vaccine — Participants will indicate which vaccine they wish to receive (Hepatitis B, Hepatitis A, or Human Papillomavirus vaccine) if they are randomized to a comparator prior to randomization.
  Arms: Group 2: Comparator
Biological: Hepatitis A vaccine — Participants will indicate which vaccine they wish to receive (Hepatitis B, Hepatitis A, or Human Papillomavirus vaccine) if they are randomized to a comparator prior to randomization.
  Arms: Group 2: Comparator
Biological: Human Papillomavirus vaccine — Participants will indicate which vaccine they wish to receive (Hepatitis B, Hepatitis A, or Human Papillomavirus vaccine) if they are randomized to a comparator prior to randomization.
  Arms: Group 2: Comparator

SUMMARY:
This is a single-centered trial of a group A streptococcal (GAS) vaccine, StreptAnova™. The study is designed to assess safety and immunogenicity of three doses (0, 1, 6 months) of one dosage (600 µg protein) in healthy adults 18 through 50 years of age.

DETAILED DESCRIPTION:
This is a single-centered trial of a group A streptococcal (GAS) vaccine, StreptAnova™, to be performed in Canada. It will be randomized, observer-blinded, and comparator controlled. The study is designed to assess safety and immunogenicity of three doses (0, 1, 6 months) of one dosage (600 µg protein) in healthy adults 18 through 50 years of age.

A comparator vaccine is included at 2:1 ratio (StreptAnova™ to comparator). Assignment to StreptAnova™ or comparator vaccine will be both randomized and observer-blinded. Three (3) 0.6 mL doses (600 µg protein) of StreptAnova™ or 0.5 mL doses of comparator will be administered on days 0, 30 and 180 (N= 30 StreptAnova™, 15 comparator); each subject will receive three doses of the same treatment.

Forty-five subjects will be enrolled. At each vaccine dose, detailed safety data will be collected from the first 15 randomized subjects until seven days after administration and used to determine whether to proceed to immunizing the 30 remaining subjects. Detailed safety data will be collected from the remaining 30 randomized subjects until seven days after administration and used to determine whether to proceed to immunizing the first 15 randomized subjects at the next dose.

Treatments will be followed by standard clinical parameters for evaluating the safety of a biologic/vaccine product including standardized methods for local and systemic vaccine reactions, repeated vital signs and physical examinations, 12-month follow-up (6 months post-dose 3) for adverse events and concomitant medication changes, and monitoring of clinical laboratory values as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy adults ages 18 to 50 years inclusive;
* Good general health as determined by screening evaluation no greater than 42 days before the first immunization;
* For women of childbearing age, use of adequate birth control from enrollment until 180 days after the last injection;
* Written informed consent, after reading the consent form and having adequate opportunity to discuss the study with an investigator or a qualified designee.

Exclusion Criteria:

* Presence of any febrile illness or any known or suspected acute illness on the day of any first immunization;
* Any chronic illness, whether or not active treatment is required;
* Any immunodeficiency (congenital or acquired);
* Any history of cardiac pathology (acquired or severe/persistent congenital);
* Any history of congenital malformation syndromes associated with congenital heart disease (syndrome complexes, e.g. VATER association; chromosomal disorders, e.g. Down's Syndrome; teratogenic agents, e.g. fetal alcohol syndrome; others, e.g. Noonan's);
* Any history of clinical manifestations of auto-immune or systemic diseases (inflammatory disorders, e.g. JRA, SLE, Kawasaki disease; inborn errors of metabolism, e.g. Fabry; connective tissue disorders, e.g. Marfan syndrome; neuromuscular disorders, e.g. Friedreich ataxia; endocrine-metabolic disorders, e.g. hypothyroidism; hematologic disorders, e.g. sickle cell anemia);
* Any history of acute rheumatic fever (ARF), post-streptococcal glomerulonephritis (PSGN), undiagnosed acute self-limiting polyarthritis (swelling, heat, redness or tenderness or pain and limitation of motion in >2 joints), or chorea (purposeless, involuntary rapid movements of the trunk and/or extremities);
* Any previous echocardiogram suggestive of cardiac pathology;
* Any immediate family history (parents, siblings) of ARF, PSGN, self-limiting polyarthritis, chorea, or a collagen-vascular disease such as Lupus or Sjögren's syndrome;
* Receipt of systemic glucocorticoids (a dose ≥ 20 mg/day prednisone or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within six months;
* Receipt of any investigational drug within six months, or prior participation in a clinical trial of a group A streptococcal vaccine;
* Receipt of blood products or immunoglobulin (IVIg or IMIg) within three (3) months of study entry/baseline serologic evaluation;
* Any physical findings suggestive of acute or chronic illness;
* History of receiving Adriamycin or other chemotherapy;
* Use of any of the following diet pills: fenfluramine, phentermine, or dexfenfluramins (also known as Pondimin, Redux, Adipex, or Fastin);
* History of sensitivity to any component of study vaccines;
* Evidence of tissue cross-reactive antibodies to human heart, joint cartilage, kidney, cerebral cortex or basal ganglia by indirect fluorescent antibody assay at pre-vaccination screening;
* Repeatable clinical laboratory abnormalities (blood or urine), as defined by lab normal ranges. To exclude transient abnormalities, the investigator may repeat a test up to twice, and if the repeat test is normal, subject may be enrolled;
* Echocardiographic finding of valvular dysfunction (stenosis, leaflet thickening or nodules, restricted leaflet mobility, or prolapse), LV dysfunction, atrial or ventricular enlargement, mild or greater mitral regurgitation or aortic insufficiency, moderate or greater tricuspid regurgitation or pulmonic insufficiency, pericardial effusion, or other cardiac pathology as identified by echocardiologist*;
* Receipt of any vaccines within 2 weeks of Dose 1;
* Clinically significant abnormality on screening electrocardiogram*
* Pregnancy or breastfeeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | Injection to Day 360, 6 months post dose 3

SECONDARY OUTCOMES:
Occurrence of any hematological and biochemical laboratory abnormality | Screening, day 0, day 7, day 30, day 44, day 180 and day 194
Occurrence of any unsolicited AE | During 28-day follow-up period after injection (i.e. the day of injection and 27 subsequent days), and through to day 360.
Serum antibodies against M protein and Spa antigens in the vaccine measured by ELISA | Visit 2 (day 0, pre dose 1), Visit 4 (day 30, 30 days post dose 1), Visit 5 (day 44, 14 days post dose 2), Visit 8 (day 210, 30 days post dose 3) and Visit 10 (day 360, 6 months post dose 3)
Functional opsonophagocytosis antibody determination for a subset of M protein serotypes | Visit 2 (day 0, pre dose 1), Visit 8 (day 210, 30 days post dose 3) and Visit 9 (day 280, 100 days post dose 3).

CONTACTS AND LOCATIONS:
Overall Officials: Shelly McNeil, MD, Principal Investigator — Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Finn MB, Penfound TA, Salehi S, Ogega CO, Dold C, Plante O, Dale JB. Immunogenicity of a 30-valent M protein mRNA group A Streptococcus vaccine. Vaccine. 2024 Sep 17;42(22):126205. doi: 10.1016/j.vaccine.2024.126205. Epub 2024 Aug 13. PMID 39141987
- [Derived] Pastural E, McNeil SA, MacKinnon-Cameron D, Ye L, Langley JM, Stewart R, Martin LH, Hurley GJ, Salehi S, Penfound TA, Halperin S, Dale JB. Safety and immunogenicity of a 30-valent M protein-based group a streptococcal vaccine in healthy adult volunteers: A randomized, controlled phase I study. Vaccine. 2020 Feb 5;38(6):1384-1392. doi: 10.1016/j.vaccine.2019.12.005. Epub 2019 Dec 13. PMID 31843270